CLINICAL TRIAL: NCT07346625
Title: Impact of Comorbiditries and Disease Severity on Clinical Outcomes of Patients With Acute Exacerbations of Bronchiectesis
Brief Title: Impact of Comorbidities and Severity on Outcomes in Bronchiectasis Excerbations
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aliaa Elsayed Mahmoud, Impact of comorbiditries and Disease severity on clinical outcomes of patients with acute exacerbations of bronchiectesis, Sohag University
Other Study IDs: Soh-Med-25-9-16MS
Record Dates: First submitted 2025-11-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis With Acute Exacerbation
MeSH Terms: interventions — Patient Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult bronchiectasis patient with acute excerbations: Group 1: Mild-to-Moderate Disease Severity Patients diagnosed with bronchiectasis who present with acute exacerbations and have mild to moderate disease severity scores (based on BSI or FACED scoring). Data on comorbidities, clinical outcomes, and hospital stay will be recorded.
  Group 2: Severe Disease Severity Patients with acute exacerbations of bronchiectasis classified as severe according to BSI or FACED score. These patients are expected to have higher comorbidity burden and worse clinical outcomes.
  Alternative grouping (if by comorbidity burden):
  Group A: With Significant Comorbidities Patients with one or more major comorbidities such as COPD, diabetes, or cardiovascular disease.
  Group B: Without Significant Comorbidities Patients without major comorbid conditions, serving as a comparison group.
  Interventions: Other: Observational assessment of comorbidities and disease severity

INTERVENTIONS:
Other: Observational assessment of comorbidities and disease severity — > This study involves no active intervention. Data will be collected from patients with acute exacerbations of bronchiectasis to assess the impact of comorbidities and disease severity on clinical outcomes such as hospital stay, ICU admission, and mortality.

SUMMARY:
Acute exacerbations of bronchiectasis are associated with variable outcomes depending on patient factors. Comorbidities such as COPD, diabetes, and cardiovascular disease, as well as disease severity scores, significantly influence hospitalization rates, length of stay, need for intensive care, and mortality. Understanding these associations helps in risk stratification, guiding management, and improving prognosis in affected patients.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic respiratory condition characterized by permanent and abnormal dilatation of the bronchi, often associated with recurrent infections, impaired mucociliary clearance, and progressive lung damage. Acute exacerbations represent a major clinical problem, contributing to significant morbidity, reduced quality of life, and increased healthcare burden.

The clinical outcomes of patients experiencing acute exacerbations of bronchiectasis are not uniform, and multiple factors influence their prognosis. Among these, comorbidities and disease severity play crucial roles. Comorbidities such as chronic obstructive pulmonary disease (COPD), asthma, cardiovascular diseases, diabetes mellitus, and chronic renal impairment can increase susceptibility to exacerbations and worsen their clinical course. The presence of these comorbid conditions is often linked to prolonged hospital stays, higher rates of intensive care admission, frequent readmissions, and increased mortality.

Similarly, the severity of underlying bronchiectasis, often assessed through validated scoring systems (e.g., Bronchiectasis Severity Index [BSI], FACED score), is strongly correlated with outcomes during exacerbations. Patients with more severe disease tend to experience more frequent and severe exacerbations, impaired lung function, greater need for intravenous antibiotics, and higher risk of complications.

Therefore, assessing both comorbidity burden and disease severity is critical in predicting outcomes, guiding clinical decision-making, and tailoring individualized management strategies for patients presenting with acute exacerbations of bronchiectasis. A comprehensive understanding of these relationships will aid in early risk stratification, optimization of treatment, and potentially reduction of adverse outcomes in this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) admitted with a diagnosis of "Bronchiectasis with acute exacerbation". The bronchiectasis exacerbation is diagnosed based on deterioration in three or more of the following main symptoms for 48h at least: cough, sputum volume or sputum consistency, purulent sputum, breathlessness or exercise tolerance, fatigue or malaise, hemoptysis, and the requirement of a change in the bronchiectasis treatment as determined by a clinician.

Exclusion Criteria:

* Patients younger than 18 years of age. Patients who refuse participation or whose medical records lack informed consent (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients (≥18 years) diagnosed with bronchiectasis who are admitted to the hospital with acute exacerbations. Patients will be recruited from the Department of Chest Diseases at Sohag University Hospital (or your hospital name). All eligible patients during the study period will be included consecutively. Data regarding demographic characteristics, comorbidities, disease severity scores (BSI or FACED), and clinical outcomes will be collected and analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical treatment failure during Bronchiectasis Exacerbation | 30 days after exacerbation onset
  composite clinical treatment failure,defined as the occurrence of any of the following events within 30 days of bronchiectasis exacerbation onset: 1.hospitalization related to the exacerbation 2.escalation or change of antibiotic therapy 3.Admission to the intensive care unit 4.Death from any cause

SECONDARY OUTCOMES:
correlation between disease severity and clinical treatment failure | 1 year
  correlation between baseline bronchiectasis severity ,assessed using the bronchiectasis severity index(BSI), and clinical treatment failure during exacerbations.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The collected data will be used only for the current study purposes and will remain confidential according to institutional regulations.